CLINICAL TRIAL: NCT03486600
Title: Safety of Fluid Resuscitation With Hydroxyethyl Starch 130/0.4 on Blood Coagulation and Renal Functions in Trauma Patients: Multicenter Clinical Trial
Brief Title: Fluid Resuscitation With Hydroxyethyl Starch 130/0.4 in Trauma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sherif M. S. Mowafy, principl investigator, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 4410/11-3-2018
Record Dates: First submitted 2018-03-12; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Trauma patients of both sexes and diagnosed to be in hemorrhagic shock and there is an expected delay in blood and blood products transfusion for more than 40 minutes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fluid resuscitation (Other): Patients will be evaluated and the bleeding site to be investigated and hemorrhagic shock confirmed and there is an expected delay in blood and blood products transfusion for more than 40 minutes. 6% HES 130/0.4 (Voluven®) will be administered intravenously to maintain or restore hemodynamic stability up to a maximum dose of 50 mL/kg body weight.
  Interventions: Other: Fluid Resuscitation

INTERVENTIONS:
Other: Fluid Resuscitation — Patients will be evaluated and the bleeding site to be investigated and hemorrhagic shock confirmed and there is an expected delay in blood and blood products transfusion for more than 40 minutes. 6% HES 130/0.4 (Voluven®) will be administered intravenously to maintain or restore hemodynamic stability up to a maximum dose of 50 mL/kg body weight.

SUMMARY:
Fluid therapy in trauma patients is considered one of the common challenges in daily practice. Both crystalloids and colloids can be used to maintain adequate blood volume and tissue perfusion but there is an ongoing debate as both of them could affect coagulation and renal function. The latest generation of the commercially available Hydroxy Ethyl Starch (HES) solutions was developed to improve pharmacokinetics and safety profile of HES, minimizing adverse effects such as impairment of blood coagulation or renal function. But data on early fluid resuscitation in trauma patients with these starches are limited and its safety on coagulation and renal function is still questioned.

DETAILED DESCRIPTION:
Fluid resuscitation is a fundamental of the initial management and resuscitation of trauma patients to preserve or restore normovolemia, cardiac output, tissue perfusion, and correcting coagulopathy and acid-base balance during massive blood loss, yet fluid therapy in trauma patients is considered one of the common challenges in our daily practice with a lot of controversies and recommendations changing from using crystalloids, colloids, and/or packed red blood cells. Also, fluid availability which does not necessarily matches the best fluid needed for the patient impacts the physician choice of fluids especially when blood is not available.Both crystalloids and colloids can be used to maintain adequate blood volume and tissue perfusion. But both of them could affect coagulation and renal function. Both crystalloids and colloids decrease concentration of coagulation factors and number of platelets causing dilutional coagulopathy. Moreover, synthetic colloids impair polymerization of fibrin and platelet function, aggravating coagulopathic state. So, their use may therefore increase blood loss. As, all hydroxyethyl starch (HES) colloid solutions are excreted through the kidneys and other ways of excretion are negligible a lot of clinical trials have raised concerns about the renal safety of HES due to observed high frequency of acute kidney injury and high mortality rates in critically ill patients.These effects depend on the pharmacokinetic properties of the HES used, which determines the HES plasma concentrations over time, in vivo molecular weight (Mw), and maximum doses used. The latest generation of the commercially available HES solutions the medium-Mw starch, HES 130/0.4 (6%, Voluven®), was developed to improve pharmacokinetics and to improve the safety profile of HES, minimizing adverse effects such as impairment of blood coagulation or renal function.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients in hemorrhagic shock
* Expected delay in blood and blood products transfusion for more than 40 minutes.

Exclusion Criteria:

* Known chronic renal disease
* Known chronic liver disease
* Known coagulopathy
* Known allergy to Hydroxyethyl starch
* Known pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 392 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Abnormal Coagulation Profile | 7 days
  abnormal coagulation profile as indicated by prothrobin time, partial thromboplastin time, international standardization ratio, prothrombin concentration and fibrengen level. Samples were collected on day one after patient stabilization.
Development of acute kidney injury | 7 days
  acute kidney injury as defined by the RIFLE (Risk, Injury, Failure, Loss, End stage kidney disease) criteria depending on serum creatinine and urine output

SECONDARY OUTCOMES:
Length of stay in the intensive care unit (ICU) | 30 days
  early fluid resuscitation with HES 130/0.4 may affect the length of stay in ICU
30-day mortality | 30 days
  the effect of HES 130/0.4 resuscitation on patient mortality
length of stay in the hospital. | 30 days
  early fluid resuscitation with HES 130/0.4 may affect the length of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Hany V Zaki, MD, Study Director — Anesthesia and Surgical Intensive Care Department, Faculty of Medicine -Ain Shams University; Sherif MS Mowafy, MD, Principal Investigator — Anesthesia and Surgical Intensive Care Department, faculty of medicine, Zagazig University; Nasr MA SeifElnasr, MD, Principal Investigator — Anesthesia and Surgical intensive care Department, Faculty of Medicine - Cairo University; Ahmed H Bakeer, MD, Principal Investigator — Anesthesia and pain relief Department, National Cancer Institute - Cairo University

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will be available 6 months after publication
Access Criteria: by contacting the study director

REFERENCES:
- [Background] Wise R, Faurie M, Malbrain MLNG, Hodgson E. Strategies for Intravenous Fluid Resuscitation in Trauma Patients. World J Surg. 2017 May;41(5):1170-1183. doi: 10.1007/s00268-016-3865-7. PMID 28058475
- [Background] (2) Jabaley C and Dudaryk R: Fluid Resuscitation for Trauma Patients: Crystalloids Versus Colloids. CurrAnesthesiol Rep 2014; 4:216-224.
- [Background] Rossaint R, Bouillon B, Cerny V, Coats TJ, Duranteau J, Fernandez-Mondejar E, Filipescu D, Hunt BJ, Komadina R, Nardi G, Neugebauer EA, Ozier Y, Riddez L, Schultz A, Vincent JL, Spahn DR. The European guideline on management of major bleeding and coagulopathy following trauma: fourth edition. Crit Care. 2016 Apr 12;20:100. doi: 10.1186/s13054-016-1265-x. PMID 27072503
- [Background] James MF, Michell WL, Joubert IA, Nicol AJ, Navsaria PH, Gillespie RS. Resuscitation with hydroxyethyl starch improves renal function and lactate clearance in penetrating trauma in a randomized controlled study: the FIRST trial (Fluids in Resuscitation of Severe Trauma). Br J Anaesth. 2011 Nov;107(5):693-702. doi: 10.1093/bja/aer229. Epub 2011 Aug 19. PMID 21857015
- [Background] Ding X, Cheng Z, Qian Q. Intravenous Fluids and Acute Kidney Injury. Blood Purif. 2017;43(1-3):163-172. doi: 10.1159/000452702. Epub 2017 Jan 24. PMID 28114128
- [Background] Masoumi K, Forouzan A, Darian AA, Rafaty Navaii A. Comparison of the Effectiveness of Hydroxyethyl Starch (Voluven) Solution With Normal Saline in Hemorrhagic Shock Treatment in Trauma. J Clin Med Res. 2016 Nov;8(11):815-818. doi: 10.14740/jocmr2702w. Epub 2016 Sep 29. PMID 27738483